CLINICAL TRIAL: NCT00005671
Title: Quality of Life in Chronic Ischemic Heart Disease With Left Ventricular Dysfunction
Brief Title: Quality of Life in Patients With Chronic Ischemic Heart Disease
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000131; 00-CC-0131
Record Dates: First submitted 2000-05-24; First posted 2000-05-25 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-05

CONDITIONS: Ischemic Heart Disease; Myocardial Ischemia
Keywords: Angina; Condition Specific; Heart Failure; Symptom Distress; Revascularization; Coronary Artery Disease; Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Heart Failure; Coronary Artery Disease

SUMMARY:
This study will examine the health-related quality of life in patients being treated for chronic heart disease.

Patients 18 years or older with chronic ischemic heart disease and left ventricular dysfunction enrolled in protocols in the National Heart Lung and Blood Institute's Cardiology Branch may participate in this study.

Participants will complete five questionnaires at 3 separate times during the study-once during hospitalization at the NIH Clinical Center and again at home 6 months and 1 year later. The questionnaires, described below, require a total of about 30 minutes to complete.

1. Demographic Information Sheet -General information such as age, marital status, employment, education, and history of cardiac medical procedures.
2. General Health Survey -Patient's self-assessment, on a rating scale, of physical and emotional well being. Questions are related to the ability to perform work and daily living activities, mood and state of mind, limitations on social activities, energy level, pain level, general quality of life, etc.
3. Heart Disease Survey - Patient's self-assessment, on a rating scale, of the level of physical, social, emotional and functional well being related to his or her heart condition. Questions concern fatigue level, emotional outlook, social well being, etc.
4. Angina Survey - Information on the frequency of chest pain, chest tightness, or angina.
5. Symptom Distress Survey - Patient's ranking of the degree of symptom distress from chest discomfort, difficulty breathing, heart rate irregularities, wheezing and coughing.

All information provided in the questionnaires will be kept confidential. Upon request, patients will be sent a summary of the study results when the study is completed.

DETAILED DESCRIPTION:
A majority of the research in patients with chronic ischemic heart disease and left ventricular dysfunction deals with increasing patient survival rates and years. Very little research has focused on patients' perceptions of living with this chronic debilitating disease. The purpose of this naturalistic, prospective study is to assess the Health Related Quality of Life (HRQOL), anginal symptoms and symptom distress experienced by patients with chronic ischemic heart disease and left ventricular dysfunction. The relationship between underlying cardiac condition, anginal symptoms, symptom distress and HRQOL will be examined. The trend in HRQOL across time versus treatment group will be evaluated. The question, does HRQOL, anginal frequency and symptom distress at baseline predict mortality and cardiac related hospitalization during the year following assessment will also be addressed.

Patients who are enrolled in protocols in the Cardiology Branch of the National Heart Lung and Blood Institute (NHLBI) and diagnosed with chronic ischemic heart disease and left ventricular dysfunction will be asked to participate in this HRQOL study. Patients will complete measures of HRQOL (Medical Outcomes Short Form 36 Survey; Minnesota Living with Heart Failure Questionnaire) and symptom measures (anginal frequency subscale of the Seattle Angina Questionnaire; cardiopulmonary subscale of the Heart Transplant Symptom Checklist). Underlying cardiac condition will be assessed using exercise thallium imaging parameters (METS and perfusion defects) and positron emission tomography (PET) imaging parameter (viability). A sample size of 90 subjects is desired for this study. Data will be analyzed using multivariate statistics. It is expected that this study will provide new information regarding how patients with ischemic heart disease and left ventricular function feel their chronic illness and its corresponding treatment(s) affects their HRQOL.

ELIGIBILITY:
Known coronary artery disease.

Left ventricular ejection fraction less that or equal to 45%.

Signed informed consent.

Must be able to read written English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105
Dates: Start 2000-05; Study Completion 2002-05

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lukkarinen H. Quality of life in coronary artery disease. Nurs Res. 1998 Nov-Dec;47(6):337-43. doi: 10.1097/00006199-199811000-00007. PMID 9835489
- [Background] Konstam V, Salem D, Pouleur H, Kostis J, Gorkin L, Shumaker S, Mottard I, Woods P, Konstam MA, Yusuf S. Baseline quality of life as a predictor of mortality and hospitalization in 5,025 patients with congestive heart failure. SOLVD Investigations. Studies of Left Ventricular Dysfunction Investigators. Am J Cardiol. 1996 Oct 15;78(8):890-5. doi: 10.1016/s0002-9149(96)00463-8. PMID 8888661
- [Background] Grady KL, Jalowiec A, Grusk BB, White-Williams C, Robinson JA. Symptom distress in cardiac transplant candidates. Heart Lung. 1992 Sep-Oct;21(5):434-9. PMID 1399662